CLINICAL TRIAL: NCT02237664
Title: Patient-Controlled Thoracic Paravertebral Block for Postoperative Analgesia After Video-Assisted Thoracoscopic Surgery
Brief Title: Patient-Controlled Thoracic Paravertebral Block After Video-Assisted Thoracoscopic Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UD-2015-16-P1Anesth; GPAnesth-1 (Other: Dammam University)
Record Dates: First submitted 2014-09-08; First posted 2014-09-11 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Video-assisted Thoracoscopic Surgery
Keywords: Thoracoscopy; Patient-controlled analgesia; Paravertebral analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient-controlled paravertebral analgesia (PC-PVB) (Active Comparator): Patient-controlled paravertebral analgesia
  Interventions: Procedure: Patient-controlled paravertebral analgesia (PC-PVB)
- Continuous paravertebral analgesia (C-PVB) (Placebo Comparator): Continuous paravertebral analgesia
  Interventions: Procedure: Continuous paravertebral analgesia (C-PVB)

INTERVENTIONS:
Procedure: Continuous paravertebral analgesia (C-PVB) — Patients will receive continuous paravertebral infusion of bupivacaine 0.2% and fentanyl 2 μg mL-1 at rate of 8 mL h-1
  Arms: Continuous paravertebral analgesia (C-PVB)
Procedure: Patient-controlled paravertebral analgesia (PC-PVB) — Patients will receive background continuous paravertebral infusion of bupivacaine 0.2% and fentanyl 2 μg mL-1 at rate of 8 mL h-1 with patient demand bolus dose of 3 mL and lockout time of 15 min with a 20 mL h-1 maximum dose, irrespective of their age
  Arms: Patient-controlled paravertebral analgesia (PC-PVB)

SUMMARY:
Thoracic surgery is commonly associated with severe postoperative pain and marked impairment of respiratory function.1 Minimally invasive video-assisted thoracic surgery (VATS) is assumed to result in better quality of life and less postoperative pain compared with standard open thoracotomy, other investigators have reported comparable patient-reported physical component summary and pain scores after VATS and thoracotomy during the first 12 months after lung resection.2 That study was non-randomized and 41% of the included patients did not complete the follow-up period.2 VATS has recently been increasing in popularity as a fast-track surgery with potential enhanced recovery after surgery.

Variety of approaches exist to manage pain after thoracotomy which could attenuate post-thoracotomy pulmonary dysfunction. Epidural analgesia has been considered for many decades to be the best method of pain relief after major thoracic surgery. In previous meta-analyses,3-5 many investigators have reported that thoracic paravertebral blockade (PVB) has comparable analgesic effects to thoracic epidural analgesia (TEA) in patients undergoing thoracotomy.

Additionally, PVB has a better side-effect profile, lower rates of failed block and is associated with a reduction in pulmonary complications.3-5 This could be extended to VATS to enhance recovery after surgery owing to effective analgesia and fewer side effects.6-7

Patient-controlled analgesia (PCA) has been advocated as a favourable model for postoperative analgesia, that allows a perfect match between intensity of pain and analgesic delivery, improves the quality of analgesia and decreases the cumulative analgesic consumption. Furthermore, the introduction of patient-controlled epidural analgesia (PCEA) with background infusion during labour gave patients a sense of control over their analgesia, reduced the total dose of local anesthetic administered, and had less motor block than those who receive continuous epidural analgesia.8-9Patient-controlled epidural analgesia (PCEA) has become increasingly popular for pain control after thoracotomy.10-12 In a previous preliminary study, McElwain et al.13 have reported satisfactory analgesia after breast cancer surgery with the use of PC-PVB, using either 15-min or 30-min lockout, that study did not include a comparative arm with a continuous paravertebral infusion. Furthermore, Abou Zeid et al. have reported comparable analgesia after thoracic surgery with the use of either patient-controlled PVB had with the use of intrathecal morphine, that study was not controlled and included few patients.14

The efficacy of the patient-controlled paravertebral blockade (PC-PVB) on the quality of postoperative analgesia and pulmonary function after VATS has not yet been studied.

DETAILED DESCRIPTION:
We hypothesizes that the use of patient-controlled paravertebral blockade (PC-PVB) after VATS will be associated with lower pain scores and less pulmonary dysfunction than continuous paravertebral blockade (PVB).

Following obtaining of the Local Ethics Committee approval and informed patient consent, 62 patients, aged 18 -70 years, American Society of Anesthesiologists (ASA) physical status II-III, undergoing elective VATS using postoperative thoracic paravertebral analgesia will be included in this prospective, randomized, controlled, double-blind study.

Before operation, forced expiratory volume in 1 s (FEV1), forced vital capacity (FVC), and peak expiratory flow rate (PEFR), were measured. On the morning before surgery, the patients will be instructed in the use of the PCA pump and a VAS. The patients will be asked to rate their experienced pain using the VAS from 0 to 100 mm with 0 representing no pain and 100 representing the worst imaginable pain.

Prior to the procedure an 18 to 20 G intravenous access will be established. Patient monitors includes electrocardiograph, non-invasive blood pressure, and pulse oximeter. All patients will be premedicated with iv midazolam 0.01-0.03 mg kg-1.

Before the induction of general anesthesia, paravertebral space ipsilateral to the thoracostomy will be identified 3 cm lateral to the spinous process of T5-8 with ultrasound-guidance (USG) using a high-frequency linear array probe of a Sonosite MTurbo ultrasound machine (MicroMaxxs ultrasound system, Sonosite Inc, Bothell, WA). After the probe was placed at the level of the T5-6 interspace, the apex of the paravertebral space will be visualized as a wedge-shaped hypoechoic space surrounded by the hyperechoic line of the pleura below and the internal intercostal membrane above. An 18 G Tuohy needle (B. Braun, Germany) will be inserted in a lateral-to-medial direction using an in-plane approach and will be kept advancing until the needle tip penetrates the internal intercostal membrane.7 A 20-G epidural catheter (B. Braun, Germany) will be introduced through Tuohy needle and advanced 3 cm into the paravertebral space. After gentle aspiration, a test dose of 3 mL of bupivacaine 0.25% with epinephrine 5 µg mL-1 will be administered through the catheter. If no significant rise in heart rate or arterial pressure will be observed, a bolus of 0.3 mL kg-1 of bupivacaine 0.25% with epinephrine (5 µg mL-1), followed by continuous paravertebral infusion of bupivacaine 0.25% and fentanyl 2 µg mL-1 at 0.1 mL kg-1 h-1 intraoperatively.15

In all patients, standard monitors and state and response entropy (SE and RE, respectively, GE Healthcare, Helsinki, Finland) based-depth of anesthesia will be applied. The radial artery will be catheterized. Anesthetic technique will be standardized in all studied patients. After preoxygenation, general anesthesia will be induced with propofol 1.5-3 mg kg-1 and target-controlled infusion (TCI) of remifentanil at an effect-site concentration (Ce) of 4 ng mL-1, to achieve the SE values below 50 and the difference between RE and SE below 10. Rocuronium (0.5 mg kg-1) will be given to facilitate the endobronchial intubation with a left-double lumen endobronchial tube and the correct position of its tip will be confirmed with a fiberoptic bronchoscope.

Anaesthesia will be maintained with 0.7-1.5 minimum alveolar concentration of sevoflurane and remifentanil Ce of 2-4 ng mL-1 to maintain the SE values below 50, the difference between RE and SE below 10 and the mean arterial blood pressure (MAP) and heart rate <20% of baseline values. Rocuronium increments will be used to maintain surgical relaxation.

Two lung ventilation (TLV) will be instituted using fraction of inspired oxygen (FiO2) of 0.4 in air, tidal volume (VT) of 8 mL kg-1, inspiratory to expiratory (I: E) ratio of 1:2.5 and PEEP of 5 cm H2O, and respiratory rate will be adjusted to achieve an arterial carbon dioxide tension (PaCO2) of 4.7-6 kPa. During one-lung ventilation (OLV), the dependent lung will be ventilated with a FiO2 of 1.0, VT of 6 mL kg-1 and I: E ratio, PEEP, and respiratory rate, will be maintained as during TLV. The dependent lung will be recruited at 30-minute intervals by increasing the inspiratory pressure to 40 cmH2O for 10 seconds.

All surgical procedures will be performed by the same surgeons who will be blinded for the study group. The VATS procedure will begin with the exploration of the pleural cavity using a 30° video thoracoscopic camera through 1.5 cm single skin incision with the use of 1-3 trocars which enables the thoracoscopic instruments to move the lung.

At the end of surgery, the nondependent lung will be re-expanded, the remifentanil and sevoflurane will be discontinued after chest closure and skin closure, respectively, and the residual neuromuscular blockade will be antagonized.

During working hours of the first 48 hours, the patients will be visited by an acute pain nurse and/or a consultant anesthesiologist, who will interview each patient regarding satisfaction with postoperative analgesia. After hours, an anesthetic registrar will be available to review analgesia management. All patients will receive multimodal analgesia consisting of regular IV paracetamol (1 g four times a day) and IV lornoxicam (8 mg two times a day) for postoperative pain relief.

Breakthrough pain, defined as pain VAS > 30 mm, will be treated with a bolus of 0.1 mL kg-1 of paravertebral medication administered through the pump. No additional medication will be given if the pain VAS < 30 mm. If after 15 minutes pain VAS persists greater than 30, additional 0.1 mL kg-1 of the paravertebral medication will be given. If the patient still has a pain VAS > 30 despite breakthrough pain intervention, then the patient will be connected to PCA with intravenous morphine 1 mg, with a lockout interval of 8 minutes and a maximum 4-hourly limit of 30 mg.5

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II-III.
* Use of postoperative thoracic paravertebral analgesia

Exclusion Criteria:

* Cardiac disease
* Pulmonary disease
* Renal disease
* Hepatic disease
* Neuropsychiatric disease
* Pregnancy
* Bleeding disorder
* Severe anatomical abnormalities of the vertebral column or ribs
* Allergy to study medications
* Other contraindications to paravertebral analgesia
* Body mass index (BMI) ≥ 35 kg m-2
* Body weight less than 50 kg
* Emergency surgery
* Preoperative pain score > 70 mm on visual analogue scale (VAS)
* Drug or alcohol abuse
* Chronic pain condition requiring daily intake of analgesics
* Language or mental disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 48 hours after surgery
  Pain scores on a 100-mm-long visual analog score (VAS) at rest and on cough

SECONDARY OUTCOMES:
Hemodynamic variables | 48 hours after surgery
  Heart rate
Number of bolus demands | 48 after surgery
  The number of bolus demands
Actual number of boluses | 48 hours after surgery
  the actual number of on demand boluses of the patient-controlled analgesia received by the patient
Total volume of administered bupivacaine | 48 hours after surgery
  total volume of bupivacaine administered during the first 48 hours after surgery
Rescue analgesic requirements | 48 hours after surgery
  rescue analgesic requirements
Requirement for antiemetic medication | 48 hours after surgery
  Requirement for antiemetic medications
Overall patient satisfaction | 48 hours after surgery
  Overall patient satisfaction will be recorded on a 100-mm visual analog scale (VAS) (0 mm = completely dissatisfied, 100 mm = completely satisfied) after catheter removal.
Sedation scores | 48 hours after surgery
  Patient sedation will be assessed 4 hourly on a five-point sedation score (1, wide awake; 2, drowsy or dozing intermittently; 3, mostly sleeping but easily awakened; 4, asleep, difficulty responding to verbal commands; 5, awakened only by shaking).
Pulmonary function tests | 24 hours before surgery, 72 hours after surgery
  , forced expiratory volume in 1 s (FEV1), forced vital capacity (FVC), and peak expiratory flow rate (PEFR) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Al Jehani, MD, Principal Investigator — Chairman of Surgery Dept; Mohamed R El Tahan, MD, Study Director — Imam Abdulrahman Bin Faisal University
Locations (1):
- King Fahd Hospital of the University, Khobar, Eastern Province, Saudi Arabia